CLINICAL TRIAL: NCT02130271
Title: PET/MRI Imaging of Neuraxial Inflammation in Sciatica Patients
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Yi Zhang, MD, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2013P-002174
Record Dates: First submitted 2014-04-24; First posted 2014-05-05 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Sciatica
Keywords: Sciatica; PET scan; MRI; Inflammation; Epidural Steroid Injection (ESI)
MeSH Terms: conditions — Sciatica; Inflammation | interventions — (methyl-(11)C)N-acetyl-N-(2-methoxybenzyl)-2-phenoxy-5-pyridinamine; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A blood sample will be taken from healthy subjects only at Visit 1. The blood sample will genotyped. Genotyping will identify if the subject makes proteins that will bind the radioactive tracer.
  A blood sample will be drawn for Genotyping at Visit 2 from all subjects.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy: Healthy subjects with no pain.
  * Radioactive dye
  * PET/MRI
  * Blood draw
  Interventions: Drug: Radioactive dye; Radiation: PET/MRI; Other: Blood draw
- Sciatica: Subjects with sciatica and scheduled for an epidural steroid injection (ESI).
  * Radioactive dye
  * PET/MRI
  * Blood draw
  Interventions: Drug: Radioactive dye; Radiation: PET/MRI; Other: Blood draw

INTERVENTIONS:
Drug: Radioactive dye — The radioactive dye [11C]PBR28 will be administered through an intravenous line (IV).
  Other Names: [11C]PBR28
Radiation: PET/MRI — All subjects will undergo a simultaneous PET/MRI scan. The scan will be up to 2 hours long.
  Other Names: Integrated MR-PET 3 Tesla scanner (Siemens Biograph mMR).
Other: Blood draw — Up to 11 tablespoons of blood will be drawn through an intravenous line (IV-line) for two purposes: 1) testing for the subject's genetic affinity to the radioactive dye, and 2) testing for the presence inflammatory biomarkers.

SUMMARY:
The purpose of this study is to see if the spine shows areas of inflammation using a specific type of imaging (pictures).

DETAILED DESCRIPTION:
The purpose of this study is to determine if inflammation around the spinal nerves can be identified using a radioactive tracer [11C] PBR28 and integrated PET/MRI scan for the purpose of better treating patients who have radicular lumbar pain with epidural steroid injections.

ELIGIBILITY:
Inclusion criteria for pain subjects:

1. Subject is 18-75 years old.
2. Subject is able to give written informed consent.
3. Subject is currently diagnosed with lower extremity radicular pain regardless of specific or suspected etiologies.
4. Subject has a clear dermatomal distribution of the painful area extending to the distal lower extremities.
5. Subject reports ongoing pain intensity of 4 or greater using the visual analogue scale (VAS) during the week prior to enrollment.

Inclusion criteria for healthy subjects:

1. Subject is 18-75 years old.
2. Subject is able to give written informed consent.
3. Subject has no history of chronic back/spine pain.

Exclusion criteria for all groups:

1. Subject recently received a lumbar ESI (within 8 weeks).
2. Subject starts new NSAID medication for pain during the study.
3. Subject has predominantly axial low back pain.
4. Subject has known pain condition secondary to hip joint arthritis.
5. Subject is pregnant or breastfeeding.
6. Subject has allergy to lidocaine.
7. Subject is treated with chronic corticosteroid therapy.
8. Subject is on anticoagulation therapy (i.e. Coumadin, Plavix, or Lovenox).
9. Subject has a known bleeding disorder (i.e. hemophilia).
10. Subject has uncontrolled high blood pressure [>170/100].
11. Subject has a known heart condition.
12. Subject has known inflammatory disease (i.e. inflammatory bowel disease; ankylosing spondylitis; etc.).
13. Subject has known liver dysfunction or renal insufficiency or impaired elimination (Renal dysfunction is defined as eGFR < 60. Hepatic dysfunction is defined as LFTs ≥ 3x ULN).
14. Subject has been hospitalized recently (within one month) for a major psychiatric disorder (i.e. major depression, bipolar disorder, schizophrenia, anxiety disorder, or psychosis).
15. Subject has contraindications to MRI and PET scanning (i.e. presence of a cardiac pacemaker or pacemaker wires, metallic particles in the body, vascular clips in the head or previous neurosurgery, prosthetic heart valves, or claustrophobia).
16. Subject had research-related radiation exposure in the last 12 months.
17. Subject tests positive for use of illicit drugs, marijuana, or non-prescribed drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Subject is currently diagnosed with lower extremity radicular/sciatica pain.
  2. Healthy subjects with no pain from the local community.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2014-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Inflammation in the spine | 2 hours
  The presence of inflammation in the spine using the radioactive tracer [11C]PBR28.

SECONDARY OUTCOMES:
Pain Scores on the Visual Analog Scale (VAS) | up to 3 months
  The subject's pain score (VAS) at baseline and up to 3 months after the ESI treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Zhang, MD, PhD., Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH Center for Translational Pain Research, Boston, Massachusetts, United States

REFERENCES:
- See also: MGH Center for Translational Pain Research — http://www.massgeneral.org/translationalpainresearch/